CLINICAL TRIAL: NCT04022226
Title: A Randomized Pilot Study Examining DCEEG Characteristics in Ketamine Versus Methohexital Induction in Depressed Patients Receiving Electroconvulsive Therapy
Brief Title: EEG Characteristics in ECT
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, Jeremy Miller, Attending Psychiatrist, University of New Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 19-228
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Electroconvulsive Therapy; Direct Current Electroencephalogram; Ketamine; Spreadind Depression
MeSH Terms: interventions — Ketamine; Methohexital

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methohexital (Active Comparator): Standard of care anesthesia that does not affect slow wave characteristics
  Interventions: Drug: Methohexital
- Ketamine (Experimental): Standard of care anesthesia that suppresses slow wave characteristics
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Induction agent that suppresses infra-slow waves
  Arms: Ketamine
Drug: Methohexital — Induction agent that does not suppress infra-slow waves
  Arms: Methohexital

SUMMARY:
The investigators will be examining slow-wave characteristics in depressed patients receiving electroconvulsive therapy (ECT) using direct current electroencephalogram (dcEEG) by anesthesia induction agent.

DETAILED DESCRIPTION:
This is a pilot project using dcEEG to look at infra-slow waves in depressed patients receiving ECT randomized to ketamine or methohexital where ketamine suppresses infra-slow waves. The rationale for this project is to identify biomarkers of treatment adequacy in ECT, which could lead to decreased morbidity and mortality with the procedure and lessen the burden of depression in our patient population.

ELIGIBILITY:
Inclusion Criteria:

* Structured Clinical Interview for DSM-5 will confirm diagnosis of MDD or BPD-depressed (with or without psychotic features
* The clinical indications for ECT including treatment resistance or a need for a rapid and definitive response;
* Hamilton Depression Rating Scale 24-item (HDRS-24) > 21; and
* Age range between 18 and 65 years of age.

Exclusion Criteria:

* Defined neurological or neurodegenerative disorder (e.g., history of head injury with loss of consciousness > 5 minutes, epilepsy, Alzheimer's disease);
* Other psychiatric conditions (e.g., schizophrenia, schizoaffective disorder, bipolar disorder)
* Current drug or alcohol use disorder, except for nicotine and marijuana
* Adults unable to consent, pregnant women, prisoner
* Non-English speakers
* Patients that cannot tolerate Methohexital and Ketamine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of New Mexico Mental Health Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: An embargo of 2 years will be placed on the data after Master's Thesis is published and placed into the vault to allow for publications. Afterwards, it will be available as along as the vault is maintained.
Access Criteria: Pilot project is being done as a part of a Master's Thesis which will be uploaded to the University of New Mexico digital repository and may contain supporting information as above.
URL: https://digitalrepository.unm.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The funding cycle was cut short secondary to COVID and it was decided to analyze DCEEG Characteristics with only one arm, the Methohexital arm (standard of care). The Ketamine arm was cancelled.
Pre-assignment Details: We had initially envisioned this as a randomized trial, but due to COVID, we restricted it to a single-arm study.
Period: Overall Study
Arm/Group | Methohexital
Started | 11
Completed (Funding was delayed secondary to COVID, impacting study design and recruitment.) | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Methohexital
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Assessed for Clinical Efficacy of ECT
Description: Quick Inventory of Depressive Symptomatology (QIDS) and Self Reporting version (QIDS-SR) - Range 0 - 48 with higher number indicating worsening depression.
  Inadequate sample size due to COVID. Study was closed.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Methohexital
Number analyzed (Participants) | 11
Participants | 11

ADVERSE EVENTS:
Time Frame: No adverse outcome were reported within the 1 year timeframe.
Description: same definition
Arm/Group | Methohexital
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT04022226/Prot_SAP_000.pdf